CLINICAL TRIAL: NCT04062578
Title: Effects Provided by a Physiotherapy Treatment Preventing Lower Extremity Injuries in Female Football Players: A Controlled Clinical Trial
Brief Title: Effects Provided by a Physiotherapy Treatment Preventing Lower Extremity Injuries in Female Football Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Loreto Ferrández Laliena, Master Student, Universidad de Zaragoza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI18/383
Record Dates: First submitted 2019-08-06; First posted 2019-08-20 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Anterior Cruciate Ligament Injuries; Injuries, Knee; Prevention & Control
Keywords: Anterior Cruciate Ligament Injuries; Injuries, Knee, Female Football; Prevention & Control
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: In order to achieve the objectives of the study the investigators have chosen to conduct a controlled clinical trial. For the clinical trial they will define two intervention groups in collaboration with two women's soccer clubs: CD Oliver Urrutia and SD Huesca.
  They will carry out the physiotherapy program of lumbopelvic stabilization and strengthening of the musculature of the hip region carried out in the CD Oliver Urrutia (Zaragoza), club where the principal investigator will have a practice contract. The club will agree to implement the physiotherapy program in training with players from the Second National Division. The SD Huesca will be the control group, in which they will only perform the pre and post intervention measurements. The selected team was the first women's team of the club, which plays in group 1 of the Aragonese territorial league.
  When selecting football clubs, they will be taken into account the same profile of players and training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD Oliver (Experimental): Female first team players of the club that plays in the National Second Division league.
  Interventions: Behavioral: Physiotherapy program of lumbopelvic stabilization and strengthening of the hip region musculature
- SD Huesca (Active Comparator): Female first team players who play in the Aragonese Territorial First league
  Interventions: Behavioral: Physiotherapy program of lumbopelvic stabilization and strengthening of the hip region musculature

INTERVENTIONS:
Behavioral: Physiotherapy program of lumbopelvic stabilization and strengthening of the hip region musculature — The intervention program will begin in August, along with the 2019/2020 season, and will finish at the end of the first round (5-6 months). It will be applied to CD Oliver players in three weekly sessions: preventive force, compensatory force and physiotherapy attention. During this intervention period, the SD Huesca players, control group, continued with their usual training program. They will not implement any physiotherapy program like the designed one for the study.

SUMMARY:
Background and justification: Women's football has a percentage of knee injury of 31.8%, and the anterior cruciate ligament lesion is between 2 and 4 times higher than the male. Injury prevention programs seek to improve the control of the neuromuscular recruitment, dynamic valgus and lumbopelvic stabilization. Recently Cibulka and Bennett have proposed a new prevention theory based on the strengthening of the external abductor and hip rotator muscles. The objective of this study is to design and carry out a physiotherapy program based on the prevention of modifiable risks factors.

Design: Controlled clinical trial

Methodology: 2 groups were formed, the first or experimental integrated by the female players from football team called CD Oliver (CDO), and control, integrated by the female players of the first team SD Huesca (SDH). The investigators will carried out an initial and final evaluation in which they will be collected data on variables of injury incidence, muscle length and torque. A physiotherapy program will be implemented that will consider three areas of weekly action during training, preventive force sessions, compensatory force sessions and physiotherapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Have a valid federal license signed by the competent medical authority.
* Be part of a team registered in the federated league.
* Train 4 and a half hours a week or more.
* Compete and train in regulatory fields, with artificial grass.
* Have a staff composed of a qualified technician, registered and in possession of the corresponding validated license.
* Sign the informed consent.

Exclusion Criteria:

- Suffering a lower limb injury at the start of the study.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-09-09 (Estimated); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in the strength of hip musculature | The measures will be taken at the beginning and at the end of the study (45 minutes per player)
  Quadriceps Hamstrings internal and external hip rotators hip abductors Hip flexors Hip extensors

SECONDARY OUTCOMES:
Change in the muscle length test | The measures will be taken at the beginning and at the end of the study (45 minutes per player)
  Ely test (active and passive) Ober test (active and passive) Ake test Pake test
Injuries Incidence | through study completion, an average of 1 year
  number and type of injuries

CONTACTS AND LOCATIONS:
Overall Officials: Loreto L Ferrández Laliena, Physiotheraphy, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Loreto Ferrández Laliena, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided